CLINICAL TRIAL: NCT06737835
Title: Metabolic Insights: the Impact of F-18 FDG PET/CT in Adult Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdel-Baset Ahmed Ali Alsanory, Assisstant lecturer, Assiut University
Other Study IDs: PET/CT in adult lymphoma
Record Dates: First submitted 2024-12-01; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma
Keywords: 18 FDG PET CT; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: 18 FDG — 18 flurodeoxy glucose PET/CT

SUMMARY:
1. To assess staging accuracy of F-18 FDG PET/CT in lymphoma
2. Determine the role of F-18 FDG PET/CT in monitoring treatment response and detecting relapse or residual disease in lymphoma
3. To evaluate FDG uptake correlation with histopathological subtypes and immunophenotypes as a prognostic factor.

DETAILED DESCRIPTION:
The incidence of lymphoma in Egypt has been increasing in recent years, with a noticeable rise in both Hodgkin's and non-Hodgkin's lymphoma cases. This increase is due to better healthcare, awareness, and diagnostic advancements. Risk factors include infections, lifestyle, genetics, and immune system issues.

Lymphoma is now the fourth most prevalent cancer among Egyptian adults, accounting for approximately 8.4% of all new cancer cases annually. As the burden of lymphoma grows, it becomes essential to develop effective strategies for its diagnosis and management.

Flurodeoxyglucose F-18 (F-18 FDG) is a radiolabeled glucose analog that accumulates in metabolically active cells, such as lymphoma cells, making F-18 FDG positron emission tomography / computed tomography scan (PET/CT) highly sensitive for detecting malignant lesions. It plays a key role in staging lymphoma by assessing the extent of disease spread.

Additionally, F-18 FDG PET/CT is essential for assessing treatment response, detecting relapses early, and evaluating the prognosis of patients, offering prognostic value by evaluating residual disease and predicting recurrence. Its ability to monitor disease progression and detect recurrent lymphoma provides critical insights that guide therapeutic decisions and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patient must be older than 18 years.
* Confirmed Diagnosis of Lymphoma: Patient must have a confirmed diagnosis of lymphoma based on histopathology and immunophenotyping.

Exclusion Criteria:

* Patients with Known concomitant malignancy.
* Pregnancy: Pregnant women due to the potential risks associated with radiation exposure from the PET/CT scan.
* Severe Renal or Hepatic Impairment: Patients with significant renal or hepatic dysfunction that could affect FDG metabolism or excretion.
* Uncontrolled Diabetes: Patients with uncontrolled diabetes (blood glucose >200 mg/dL), as it can affect FDG uptake and PET/CT results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective study data collected from a single-center Clinical Oncology and Nuclear Medicine Department - Assuit University Hospital, which included 62 lymphoma cases who underwent F-18 FDG PET/CT for disease staging, treatment response assessment, or post-treatment monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
primary | 3 years
  Treatment Response Using Deauville Score for FDG Uptake Evaluation:
  Evaluate FDG uptake using the 5-point scale:
  1. No uptake above background
  2. Uptake ≤ mediastinum
  3. Uptake > mediastinum but ≤ liver
  4. Moderately increased compared to liver
  5. Markedly increased compared to liver X: New uptake, unlikely related to lymphoma

SECONDARY OUTCOMES:
secondary | 3 years
  Detect early relapse or residual disease using F-18 FDG PET/CT using SUVmax, maximum standardized uptake value(g/mL )

CONTACTS AND LOCATIONS:
Overall Officials: Esraa R Hassan, MD, Study Director — South Egypt Cancer Institute
Locations (1):
- Nuclear medicine- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided